CLINICAL TRIAL: NCT02141828
Title: A Phase 1 Dose Escalation and Expanded Cohort Study of EPZ-5676 in the Treatment of Pediatric Patients With Relapsed/Refractory Leukemias Bearing a Rearrangement of the MLL Gene
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Epizyme, Inc. (Industry)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor
Organization: Ipsen (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EPZ-5676-12-002
Record Dates: First submitted 2014-05-11; First posted 2014-05-20 (Estimated); Last update posted 2023-06-18 (Actual); Status verified 2020-05

CONDITIONS: Leukemia; Acute Myeloid Leukemia; Acute Lymphocytic Leukemia; Acute Leukemias
Keywords: Leukemia; Advanced hematologic malignancies; Epizyme; Phase 1b; MLL gene; 11q23; Ambiguous lineage; ALL; AML; Acute leukemias; MLL-r
MeSH Terms: conditions — Leukemia; Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — EPZ-5676

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- EPZ-5676 (Experimental): EPZ-5676 Dose escalation and expansion cohorts
  Interventions: Drug: EPZ-5676

INTERVENTIONS:
Drug: EPZ-5676 — 28-day continuous IV infusion of each 28-day cycle, given until disease progression or unacceptable toxicity develops.
  Other Names: EPZ5676; DOT1L

SUMMARY:
A subset of patients with acute myeloid leukemia (AML) and acute lymphoblastic leukemia (ALL) harbor rearrangements of the MLL gene, which are detected either by cytogenetic or fluorescent in situ hybridization evaluation at the time of diagnosis. A protein called DOT1L plays an important role in the malignant process in these leukemias. EPZ-5676 is a molecule that blocks the activity of DOT1L, and is therefore being evaluated in the treatment of patients with MLL-rearranged leukemias.

DETAILED DESCRIPTION:
This is a Phase 1b study of EPZ-5676 in pediatric patients. The study will have two phases. The first phase will assess escalating doses of EPZ-5676 in order to determine the maximally tolerated dose (MTD) or recommended phase 2 dose (RP2D) of EPZ-5676 as a 28-day continuous IV infusion. Once the MTD and/or RP2D is established, a second phase of the study will further evaluate the safety of EPZ-5676 and assess the anti-leukemia activity.

ELIGIBILITY:
Inclusion Criteria:

1. Age: >3 months to <18 years of age.
2. Diagnosis: Patients must have documented relapsed/refractory ALL, AML, or acute leukemia of ambiguous lineage and meet the following criteria:

   * Patients must have at least received an appropriate induction therapy regimen. Patients with persistent leukemia after induction therapy, or with recurrence of leukemia at any time during the course of treatment (including allogeneic HSCT) are eligible;
   * Patients must have > 10% leukemic blasts in the bone marrow;
   * Patients must have rearrangement involving the MLL gene, including reciprocal chromosomal translocations involving 11q23 by FISH, cytogenetic analysis, polymerase chain reaction (PCR) or next-generation sequencing (NGS) OR partial tandem duplication (PTD) of MLL by PCR or NGS.
3. Therapeutic Options: Patients must be ineligible or inappropriate for other treatment regimens known to have curative potential.
4. Performance Level: Karnofsky > 50% for pts > 12 years; Lansky > 50% for pts < 12 years of age.
5. Prior Therapy: Patients must have fully recovered from the acute toxic effects of all prior chemotherapy, immunotherapy, or radiotherapy prior to entering this study.

   Myelosuppressive Chemotherapy:
   * 14 days must have elapsed since the completion of cytotoxic therapy
   * Patients may receive hydroxyurea, low-dose cytarabine and/or glucocorticoids to control peripheral blood leukemic cell counts at study entry
   * At least 7 days since the completion of therapy with hematopoietic growth factors
   * At least 7 days since the completion of therapy with a biologic agent
   * At least 21 days since receipt of chimeric antigen receptor therapy or other modified T cell therapy
   * At least 60 days from prior total body irradiation (TBI)
   * At least 60 days must have elapsed from hematopoietic stem cell transplantation (HSCT)
6. Renal and Hepatic Function: Patient must have adequate renal and hepatic functions as indicated by the following laboratory values:

   * Patient must have a calculated creatinine clearance or radioisotope GFR > 60mL/min/1.73m2 or a normal serum creatinine based on age/gender
   * Total bilirubin < 1.5 x ULN for age or normal conjugated bilirubin
   * ALT and AST < 3 x ULN (unless attributed to leukemic involvement)
7. Cardiac Function: Patient must have a shortening fraction (SF) of > 27% or an ejection fraction (EF) of > 50% by echocardiogram or MUGA scan.

Exclusion Criteria:

1. Patients with CNS 3 disease or symptomatic CNS disease
2. Clinically active heart disease including prolonged QTc or prolonged PR interval, or history of arrhythmias
3. On immunosuppressive or other anti-leukemic therapy, excluding patients receiving glucocorticoids for management of circulating blast count or patients on a stable dose (<20mg/m2/day prednisone or equivalent) of systemic or topical glucocorticoid therapy with ≤ Grade 1 GvHD or tapering dose of calcineurin inhibitor
4. Patients with known bleeding diathesis or prothrombin time (PT) or aPTT >1.5 x ULN or fibrinogen <0.5 x LLN
5. Receiving prophylactic use of hematopoietic colony stimulating factors
6. Known history of infection with human immunodeficiency virus (HIV) or chronic infection with hepatitis B virus (HBsAg positive) or hepatitis C virus (anti-HCV positive)
7. Being actively treated for another concurrent malignancy
8. Pregnant or nursing females;
9. Male patients not willing to use a condom
10. Uncontrolled intercurrent illness including, but not limited to uncontrolled infection, significant graft-versus-host-disease (GvHD) (Grade 2-4), or psychiatric illness/social situations that would limit compliance with study requirements
11. Patients who are concurrently receiving strong inducers/inhibitors of CYP3A
12. Patients with known history of Trisomy 21 (Down Syndrome), history of congenital immunodeficiency or inherited marrow failure disorder.
13. Patients with known bleeding diathesis, or PT (Prothrombin time) or aPTT (activated partial thromboplastin time) > 1.5x ULN or <0.5x LLN.

Ages: 3 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 18 (Actual)
Dates: Start 2014-05; Primary Completion 2016-05 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Determine the maximum tolerated dose (MTD) and/or recommended phase 2 dose (RP2D) of EPZ-5676. | 12 months
  To determine the maximum tolerated dose (MTD) and/or recommended phase 2 dose (RP2D) of EPZ-5676 as determined by incidence of protocol-specified dose-limiting adverse events.
To assess the safety and tolerability of EPZ-5676 administered as a continuous intravenous (CIV) infusion | 22 months
  Safety and tolerability will be assessed by the incidence of adverse events in patients treated with EPZ-5676 and the evaluation of adverse events, vital signs, physical examination, 12-lead ECG, and laboratory assessments.

SECONDARY OUTCOMES:
Determine the pharmacokinetic (PK) and pharmacodynamic (PD) profile of EPZ-5676 | 18 months
  The pharmacokinetic (PK) profile will include the analysis of Cmax, AUC and steady state concentration of EPZ-5676.
  The pharmacodynamic (PD) profile will assess the effects of EPZ-5676 in peripheral blood mononuclear (PBMC) and bone marrow cells.
Evaluate early evidence of anti-tumor activity | 18 months
  Anti-tumor activity will be assessed by objective response (OR) in pediatric patients

OTHER OUTCOMES:
To determine cerebrospinal fluid (CSF) concentrations EPZ-5676 in pediatric patients receiving EPZ-5676 by CIV infusion | 18 months
Analysis of tumor cells for somatic mutations as potential predictors of response | 18 months
  Somatic mutations to include mRNA and proteins or markers of biological pathways as potential predictors of response to EPZ-5676 treatment

CONTACTS AND LOCATIONS:
Overall Officials: Neal Shukla, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center; Lia Gore, MD, Principal Investigator — Children's Hospital Colorado; Pat Brown, MD, Principal Investigator — Johns Hopkins University; Lewis Silverman, MD, Principal Investigator — Dana Farber; Maureen O'Brien, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati; Jim A Whitlock, MD, Principal Investigator — Hospital of Sick Kids; Cynthia Wetmore, MD PhD, Principal Investigator — Emory Children's Healthcare of Atlanta; Mignon Loh, MD, Principal Investigator — University of California, San Francisco; Paul Gaynon, MD, Principal Investigator — Children's Hospital Los Angeles; Todd Cooper, MD, Principal Investigator — Seattle Children's Hospital
Locations (9):
- United States (8):
  - Childrens Hospital Los Angeles, Los Angeles, California
  - University of California San Francisco Medical Center-Parnassus, San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Emory Children's Healthcare of Atlanta, Atlanta, Georgia
  - Johns Hopkins University, Baltimore, Maryland
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
- The Hospital for Sick Kids, Toronto, Ontario, Canada